CLINICAL TRIAL: NCT01024504
Title: A Multicenter Phase II Study of the Capecitabine, Oxaliplatin and Bevacizumab as First-line Treatment in Elderly Patients With Metastatic Colorectal Cancer
Brief Title: Capecitabine Plus Oxaliplatin Plus Bevacizumab as First-line Treatment in Elderly Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: John Souglakos, University Hospital of Crete
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/06.12
Record Dates: First submitted 2009-11-26; First posted 2009-12-02 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Cancer; Colorectal cancer; Elderly; Chemotherapy; Capecitabine; Oxaliplatin; Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Oxaliplatin; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XELOX/Avastin (Experimental): Capecitabine Oxaliplatin Bevacizumab
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin at the dose of 85 mg/m2 over a 4 hour intravenous infusion at day 1 every 2 weeks for a maximum of 12 consecutive cycles
  Other Names: Eloxatin
Drug: Capecitabine — Capecitabine at the dose of 1500 mg/m2 per os at days 1 to 7 every 2 weeks for a maximum of 12 consecutive cycles
  Other Names: Xeloda
Drug: Bevacizumab — Bevacizumab at the dose of 5 mg/Kgr (intravenous infusion) at day 1, every 2 weeks for a maximum of 12 consecutive cycles
  Other Names: Avastin

SUMMARY:
This trial will evaluate the efficacy and safety of the capecitabine and oxaliplatine plus bevacizumab combination as first-line treatment in elderly patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Capecitabine, oxaliplatin and bevacizumab are well known active agents in the treatment of mCRC. The treatment of elderly patients with mCRC is an area of investigation. The role of comprehensive geriatric assessment in treatment efficacy and tolerance is an area of investigation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum
* Stage IV
* Existence of two-dimensional measurable disease. The measurable disease should not have been irradiated.
* Absence or irradiated and stable central nervous system metastatic disease.
* Life expectancy of more than 3 months.
* Age ≥ 70 years.
* Performance status (WHO) ≤ 2.
* Adequate bone marrow function (Absolute neutrophil count >1000/mm3, Platelet count >100000/mm3, Hemoglobin >9gr/mm3).
* Adequate liver (Bilirubin <1.5 times upper limit of normal and SGOT/SGPT <2 times upper limit of normal).
* Creatinine clearance (Cockcroft-Gault formula) >30ml/min.
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer.
* Presence of a reliable care giver.
* Informed consent.

Exclusion Criteria:

* Prior chemotherapy for metastatic disease.
* History of thromboembolic disease or myocardial infraction within the last 6 months.
* Peripheral neuropathy ≥ grade 2.
* Bowel obstruction or chronic diarrhea.
* Psychiatric illness or social situation that would preclude study compliance.
* Other concurrent uncontrolled illness.
* Other concurrent investigational agents.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2006-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 2 - 4 months

SECONDARY OUTCOMES:
Toxicity profile | Toxicity assessment on each cycle
Time to tumor progression | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John Souglakos, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology; Lampros Vamvakas, MD, Principal Investigator — University Hospital of Crete
Locations (6):
- Greece (6):
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - Air Forces Military Hospital of Athens, Athens
  - IASO General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - Laikon General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - State General Hospital of Larissa, Larissa
  - Theagenion Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki

REFERENCES:
- [Derived] Vamvakas L, Matikas A, Karampeazis A, Hatzidaki D, Kakolyris S, Christophylakis C, Boukovinas I, Polyzos A, Georgoulias V, Souglakos J. Capecitabine in combination with oxaliplatin and bevacizumab (AXELOX) as 1st line treatment for fit and vulnerable elderly patients (aged >70 years) with metastatic colorectal cancer (mCRC): a multicenter phase II study of the Hellenic Oncology Research Group (HORG). BMC Cancer. 2014 Apr 22;14:277. doi: 10.1186/1471-2407-14-277. PMID 24755296